CLINICAL TRIAL: NCT07099482
Title: Effectiveness of Propolis Phonophoresis on Wound Healing in Diabetic Ulcer: a Randomized Controlled Trial
Brief Title: "Ultrasound-Enhanced Propolis Therapy for Healing Diabetic Foot Wounds"
Acronym: PEARL
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sinai University (Other)
Responsible Party: Principal Investigator, Amany Gomaa Atiaa, lecturer, Sinai University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SU.REC.2025(47H)
Record Dates: First submitted 2025-07-25; First posted 2025-08-01 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Diabetic Foot Ulcer t; Type 1 Diabetes Mellitus; Type 2 Diabetes Mellitus; Wound Management; Chronic Wound Healing
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: Two-arm, randomized, double-blind, controlled trial comparing propolis phonophoresis versus standard wound care.
Who Masked: Participant, Care Provider
Masking Description: Participants in both groups receive what appears to be the same treatment procedure. The intervention group receives active ultrasound therapy, while the control group receives a sham (non-therapeutic) ultrasound, keeping both participants and care providers blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: Propolis Phonophoresis (Experimental): Participants will receive topical application of 10% propolis gel on the diabetic foot ulcer followed by therapeutic ultrasound (phonophoresis) using 1 MHz frequency, 0.5-1.5 W/cm² intensity, pulsed mode (20%), for 5 minutes per session, 3 sessions/week for 4 weeks
  .Interventions:
  * Drug: Propolis gel (10%)
  * Device: Therapeutic ultrasound (phonophoresis)
  Interventions: Device: Sham ultrasound (placebo); Drug: Propolis gel (10%)
- Standard Wound Care + Sham Ultrasound (Placebo Comparator): Participants will receive conventional wound care including debridement, cleaning, and dressing. A sham ultrasound device that emits no therapeutic waves will be applied to simulate the intervention procedure.
  Interventions:
  * Other: Standard wound care procedures
  * Device: Sham ultrasound (placebo)
  Interventions: Device: Sham ultrasound (placebo)

INTERVENTIONS:
Device: Sham ultrasound (placebo) — Participants will receive conventional wound care including debridement, cleaning, and dressing. A sham ultrasound device that emits no therapeutic waves will be applied to simulate the intervention procedure.
  Other Names: Standard wound care procedures (placebo)
Drug: Propolis gel (10%) — Participants will receive topical application of 10% propolis gel on the diabetic foot ulcer followed by therapeutic ultrasound (phonophoresis) using 1 MHz frequency, 0.5-1.5 W/cm² intensity, pulsed mode (20%), for 5 minutes per session, 3 sessions/week for 4 weeks.
  Arms: Experimental: Propolis Phonophoresis

SUMMARY:
This study aims to evaluate whether using ultrasound (phonophoresis) can help deliver propolis-a natural compound made by bees-more effectively into the skin to speed up wound healing in people with diabetic foot ulcers. Diabetic foot ulcers are a common and serious complication of diabetes and often take a long time to heal. Propolis has natural anti-inflammatory and antimicrobial properties that may promote healing, but it does not easily penetrate the skin. By using ultrasound to enhance absorption, this study tests whether combining propolis with phonophoresis is more effective than standard wound care alone. Participants will be randomly assigned to receive either the propolis ultrasound therapy or standard care. The study will measure wound size, healing time, pain, infection rates, and quality of life.

DETAILED DESCRIPTION:
This randomized, double-blind, controlled clinical trial investigates the therapeutic effectiveness of propolis phonophoresis in treating diabetic foot ulcers (DFUs). DFUs affect approximately 25% of diabetic patients and are associated with high morbidity, prolonged healing, and significant healthcare costs. Propolis, a resinous substance produced by honeybees, has shown antimicrobial, anti-inflammatory, and wound-healing properties in previous studies. However, its limited skin permeability reduces its clinical utility when used topically.

Phonophoresis is a non-invasive technique that uses ultrasound waves to enhance transdermal drug delivery. This study combines a 10% propolis gel with therapeutic ultrasound (1 MHz, 0.5-1.5 W/cm², pulsed mode at 20%) to evaluate its impact on wound healing outcomes compared to standard wound care. The intervention group will receive propolis phonophoresis therapy three times per week for four weeks. The control group will receive standard wound care and a sham ultrasound.

Primary outcome measures include the percentage reduction in wound area, assessed via digital planimetry. Secondary outcomes include time to full wound closure, pain scores, infection rates, and quality-of-life assessments. The study is designed to explore whether this combined therapeutic approach can offer a clinically superior and non-surgical treatment alternative for patients with chronic diabetic ulcers.

ELIGIBILITY:
Inclusion Criteria:

Adults aged 18 to 75 years

Diagnosed with type 1 or type 2 diabetes mellitus

Presence of a diabetic foot ulcer classified as Grade 1 or 2 (Wagner classification)

Ulcer size between 1 cm² and 5 cm²

Able and willing to provide informed consent

Exclusion Criteria:

Severe infection or presence of osteomyelitis at the ulcer site

Use of systemic immunosuppressants or corticosteroids

Known allergy or hypersensitivity to propolis

Pregnant or breastfeeding women

Participation in another clinical trial within the past 30 days

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-09-30 (Estimated); Primary Completion 2026-08-25 (Estimated); Study Completion 2026-09-25 (Estimated)

PRIMARY OUTCOMES:
Percentage Reduction in Wound Area | Baseline to Week 4
  The primary outcome will be the percentage reduction in the surface area of the diabetic foot ulcer from baseline to the end of the 4-week treatment period. Wound size will be measured using digital planimetry based on standardized wound photographs.